CLINICAL TRIAL: NCT00604812
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability, and Single-Dose Pharmacokinetics of MK0462 in Subjects With Migraines Aged 6 to 17 Years
Brief Title: Drug Study in Pediatric Subjects With Migraines (MK0462-083 AM1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0462-083; 2007_601
Record Dates: First submitted 2007-10-17; First posted 2008-01-30 (Estimated); Results first posted 2009-09-02 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2022-02

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Panel A Rizatriptan (Experimental): Subjects allocated to Panel A and randomized to receive a single dose of rizatriptan 5 mg orally disintegrating tablet (ODT) on Day 1.
  Subjects weighing 20-39 kg were allocated to Panel A.
  Interventions: Drug: rizatriptan benzoate (5 mg)
- Panel A Placebo (Placebo Comparator): Subjects allocated to Panel A and randomized to receive a single dose of rizatriptan 5 mg orally disintegrating tablet (ODT) placebo on Day 1.
  Subjects weighing 20-39 kg were allocated to Panel A.
  Interventions: Drug: Rizatriptan 5 mg Placebo
- Panel B Rizatriptan (Experimental): Subjects allocated to Panel B and randomized to receive a single dose of rizatriptan 10 mg orally disintegrating tablet (ODT) on Day 1.
  Subjects weighing 40 kg and above were allocated to Panel B.
  Interventions: Drug: rizatriptan benzoate (10 mg)
- Panel B Placebo (Placebo Comparator): Subjects allocated to Panel B and randomized to receive a single dose of rizatriptan 10 mg orally disintegrating tablet (ODT) placebo on Day 1.
  Subjects weighing 40 kg and above were allocated to Panel B.
  Interventions: Drug: Rizatriptan 10 mg Placebo
- Panel C Rizatriptan (Experimental): Subjects allocated to Panel C and randomized to receive a single dose of rizatriptan ODT on Day 1. Subjects in Panel C weighing 20-39 kg received a 5 mg dose and subjects weighing 40 kg and above received a 10 mg dose.
  Panel C was added to the study by amendment to increase the number of male subjects in the 12-17 year old age group.
  Interventions: Drug: rizatriptan benzoate (5 mg); Drug: rizatriptan benzoate (10 mg)
- Panel C Placebo (Placebo Comparator): Subjects allocated to Panel C and randomized to receive a single dose of rizatriptan ODT placebo on Day 1. Subjects in Panel C weighing 20-39 kg received a 5 mg placebo dose and subjects weighing 40 kg and above received a 10 mg placebo dose.
  Panel C was added to the study by amendment to increase the number of male subjects in the 12-17 year old age group.
  Interventions: Drug: Rizatriptan 5 mg Placebo; Drug: Rizatriptan 10 mg Placebo

INTERVENTIONS:
Drug: rizatriptan benzoate (5 mg) — A single dose of rizatriptan 5 mg administered on Day 1.
  Other Names: MAXALT®; MK0462
  Arms: Panel A Rizatriptan; Panel C Rizatriptan
Drug: rizatriptan benzoate (10 mg) — A single dose of rizatriptan 10 mg administered on Day 1.
  Other Names: MAXALT®; MK0462
  Arms: Panel B Rizatriptan; Panel C Rizatriptan
Drug: Rizatriptan 5 mg Placebo — A single dose of rizatriptan 5 mg placebo administered on Day 1.
  Arms: Panel A Placebo; Panel C Placebo
Drug: Rizatriptan 10 mg Placebo — A single dose of rizatriptan 10 mg placebo administered on Day 1.
  Arms: Panel B Placebo; Panel C Placebo

SUMMARY:
A study to assess the safety, tolerability, and single dose pharmacokinetics of a marketed drug in pediatric subjects with migraines.

After completion of a portion of the study (Panels A and B), a regulatory agency issued an amended request that the 12-17 year old age group studied should include a similar number of male and female subjects. Therefore, the study was amended to add an additional panel of subjects (Panel C) to ensure gender balance specifically in this age group.

ELIGIBILITY:
Inclusion Criteria:

* Panel A and B: Male and female subjects (non-smokers) ages 6 to 17 with a history of migraines
* Panel C: Male subjects (non-smokers) ages 12 to 17 with a history of migraines
* Subject has a history of migraine headaches, and is not experiencing a migraine on the day of study drug administration

Exclusion Criteria:

* Subject has no history of migraine headaches
* Taking medications that are monoamine oxidase inhibitors (MAOI) and selective serotonin reuptake inhibitors (SSRI)
* Subject has a condition which, in the opinion of the investigator, may interfere with optimal participation in the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2007-12-17 (Actual); Primary Completion 2010-09-17 (Actual); Study Completion 2010-09-17 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fraser IP, Han L, Han TH, Li CC, Hreniuk D, Stoch SA, Wagner JA, Linder S, Winner P. Pharmacokinetics and tolerability of rizatriptan in pediatric migraineurs in a randomized study. Headache. 2012 Apr;52(4):625-35. doi: 10.1111/j.1526-4610.2011.02069.x. Epub 2012 Jan 30. PMID 22289113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Panel C was added to the study by amendment after enrollment of Panels A and B were completed.
Period: Overall Study
Arm/Group | Panel A Rizatriptan | Panel A Placebo | Panel B Rizatriptan | Panel B Placebo | Panel C Rizatriptan | Panel C Placebo
Started | 9 | 3 | 10 | 3 | 5 | 1
Completed | 9 | 3 | 10 | 3 | 5 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Panel A: Includes the participants from the 5 mg rizatriptan group (9) and the matching placebo group (3)
- Panel B: Includes the participants from the 10 mg rizatriptan group (10) and the matching placebo group (3)
- Panel C: Includes the participants who received 5 mg rizatriptan (n=1), 10 mg rizatriptan (n=4), and the matching placebo (n=1)
- Total: Total of all reporting groups
Arm/Group | Panel A | Panel B | Panel C | Total
Number analyzed (Participants) | 12 | 13 | 6 | 31
Age, Customized [Number; unit: years]
  Ages 6 to <12 | 11 (1.44) | 2 (2.14) | 0 | 13
  Ages 12 to 17 | 1 | 11 | 6 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 0 | 13
  Male | 7 | 5 | 6 | 18
Weight [Number; unit: participants]
  20-39 kg | 12 | 0 | 1 | 13
  ≥ 40 kg | 0 | 13 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Single Doses of Rizatriptan in Pediatric Migraineurs
Description: All adverse experiences spontaneously reported by subject and/or observed by investigator and repeated clinical evaluation of physical examinations, vital signs, 12-lead ECG (electrocardiogram) and laboratory safety tests (hematology/blood chemistry/urinalysis)
Time Frame: 24 Hours
Population: All Subjects as Treated- All subjects who received at least one dose of the investigational drug was used for assessments of safety and tolerability.
Measure: Number; unit: Participants
Groups:
- Rizatriptan 5 mg: Combined subjects from Panel A and Panel C randomized to receive a single dose of rizatriptan 5 mg orally disintegrating tablet (ODT) on Day 1.
- Rizatriptan 10 mg: Combined subjects from Panel B and Panel C randomized to receive a single dose of rizatriptan 10 mg orally disintegrating tablet (ODT) on Day 1.
- Placebo: Combined Placebo groups from panels A, B, and C.
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Placebo
Number analyzed (Participants) | 10 | 14 | 7
Participants
  Serious Adverse Events | 0 | 0 | 0
  Non-Serious Adverse Events | 3 | 7 | 3
  No Adverse Events Reported | 7 | 7 | 4

2. Secondary Outcome: Preliminary Pharmacokinetic Data Following Single Dose Administration of Rizatriptan- Area Under the Curve (AUC(0-∞))
Description: Preliminary pharmacokinetics data; Area Under the Curve (AUC(0-∞)); i.e., area under the concentration-time plot
Time Frame: 24 Hours
Population: Per Protocol-The set of data generated by the subset of subjects who comply with the protocol sufficiently to ensure that these data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance covers exposure to treatment, availability of measurements and absence of major protocol violations.
Measure: Mean (Standard Deviation); unit: ng hr/mL
Arm/Group | Panel A Rizatriptan | Panel B Rizatriptan | Panel C Rizatriptan
Number analyzed (Participants) | 9 | 10 | 5
ng hr/mL | 59.4 (11.5) | 84.0 (19.8) | 67.93 (25.17)

3. Secondary Outcome: Preliminary Pharmacokinetic Data Following Single Dose Administration of Rizatriptan - Maximum Concentration (Cmax)
Description: Preliminary pharmacokinetics data; Maximum concentration (Cmax); i.e, highest concentration of drug achieved
Time Frame: 24 Hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panel A Rizatriptan | Panel B Rizatriptan | Panel C Rizatriptan
Number analyzed (Participants) | 9 | 10 | 5
ng/mL | 24.6 (7.2) | 25.0 (8.1) | 18.4 (5.5)

4. Secondary Outcome: Preliminary Pharmacokinetic Data Following Single Dose Administration of Rizatriptan - Time to Maximum Concentration (Tmax)
Description: Preliminary pharmacokinetics data; Time to maximum concentration (Tmax); i.e., amount of time required to reach maximum concentration
Time Frame: 24 Hours
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Panel A Rizatriptan | Panel B Rizatriptan | Panel C Rizatriptan
Number analyzed (Participants) | 9 | 10 | 5
Hours | 1.0 [0.3 to 2.0] | 1.5 [0.3 to 3.0] | 1.3 [0.7 to 1.7]

5. Secondary Outcome: Preliminary Pharmacokinetic Data Following Single Dose Administration of Rizatriptan - Apparent Half-life (Apparent t½)
Description: Preliminary pharmacokinetics data; Apparent half-life (t½)
Time Frame: 24 Hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Panel A Rizatriptan | Panel B Rizatriptan | Panel C Rizatriptan
Number analyzed (Participants) | 9 | 10 | 5
Hours | 1.3 (0.1) | 1.6 (0.2) | 1.6 (0.4)

ADVERSE EVENTS:
Arm/Group | Rizatriptan 5 mg | Rizatriptan 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/14 | 0/7
Other Adverse Events (participants affected / at risk) | 3/10 | 7/14 | 3/7
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rizatriptan 5 mg (N=10) | Rizatriptan 10 mg (N=14) | Placebo (N=7)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Bruising of arm (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Earache (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Visual disturbance (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Tiredenss (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cold (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Painful left arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Elevation in blood pressure (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Pharmacokinetic data presented are preliminary data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.